CLINICAL TRIAL: NCT02702531
Title: Prospective, Randomized Comparison of the Use of FloShield Air System ® Versus the Referenced Technic (Water + Povidone-Iodine Solution) During Gynecologic Endoscopic Surgery to Evaluate the Operative Lens Vision Quality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tenon Hospital, Paris (Other)
Responsible Party: Principal Investigator, Pr. Emile Darai, MD, PhD, Tenon Hospital, Paris
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A01421-48
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: The Performance Evaluations of the FloShield Defogging and Cleaning System
Keywords: Laparoscopic Surgery; FloShield Defogging and Cleaning System; Clearify Defogging and Cleaning System; gynecologic

ARMS (2):
- FloShield (Experimental): FloShield Air Laparoscopic Cleaning and Defogging System used during laparoscopic surgery
  Interventions: Device: FloShield Defogging and Cleaning System
- Water + Povidone-iodine Solution (Experimental): Clearify Visualization with Water + Povidone-iodine Solutionused during laparoscopic surgery
  Interventions: Device: FloShield Defogging and Cleaning System

INTERVENTIONS:
Device: FloShield Defogging and Cleaning System

SUMMARY:
Endoscopic surgical procedures are becoming more common in all surgical specialties including gynecology that was one of the pioneers in this field specialties.

Maintaining a quality field of view is important not only to patient safety but also for the quality of surgery and reduced surgery time.

The lenses of vision which are located at the distal end of the optical vision are during endoscopic surgery in direct contact with the anatomical structures. These lenses are found soiled by several phenomena whose appearance of a mist which constitutes a major obstacle to a clear field.

The alteration of the vision requires the surgeon extraction optics in order to achieve a cleaning of the lens. This cleaning is carried out as many times as necessary. Many strategies have been developed to improve the quality of vision. These methods relate to both the development of new optical vision but also the development of the lens cleaning material. In practice, the cleaning is carried out using a sterile swab sterile saline associated with the betadine iodine.

Recently a new material called "FloShield Air System Vision System" has been proposed and has the particularity to combine both anti-fog product and a temperature control system in contact with the lens in order to fight against condensation and smoke. The purpose of this is to improve the quality of vision by reducing the fogging phenomenon and no change of the temperature in contact with the lens (moisture reduction). Accordingly, it is assumed a reduction in the number of stay and a reduction in the specific operative time associated with this cleaning.

In this context, we wish to evaluate the effectiveness of FloShield Air System vision system on the basis of a comparative, prospective, randomized against the reference method (sterile water solution + Betadine) during endoscopic surgery gynecology.

DETAILED DESCRIPTION:
The reduction in vision during endoscopic surgery is a common problem for all surgical specialties and recurring. Studies of the pathophysiological mechanisms explaining the visual impairment by fogging emphasize the role of intraperitoneal temperature and moisture in contact with the optical lens. To this can be added two other causes of impaired vision are fluid projections and passively encountered tissues during exploration (eg, blood, fat, and ascites) and products of reactions of tissue during surgery for example, the outcome of smoke using coagulation material or section. In these situations the vision may be impaired in critical times during which an optimal view is needed to improve the quality of surgery.

A report by the World Health Organization was intended to identify the consequences of impaired vision during laparoscopic surgery. It is emphasized that impaired vision can contribute to surgical errors such as the use of a device incorrectly or displacement of the instruments on structures other than those intended. Moreover, it is reported an increase in the operative time associated with suboptimal view. Finally, the psychological dimension on the disruption of the surgeon is raised with a risk of difficulty of the procedure. To minimize these problems anti mist vision solutions combined with condensed water vapor spray system are among others marketed in recent years.

The action mechanism of these systems is to distribute steam droplets condensed on the surface of the cold lens to improve the quality of vision. Most, however, require cleaning of optics, but with less theoretical frequency. Although their use is reported in the literature their use has never been evaluated on the basis of a robust methodology.

Alternative methods readily available such as povidone iodine act similarly and are significantly less expensive (at least 10 times) than the above mentioned materials. No comparative study is currently available to support the effectiveness of these materials to the reference method inexpensive but partially effective. Their use is based solely on experience and expert opinion.

Vision device "FloShield Air System" was developed. We offer a comparative evaluation of the effectiveness of FloShield Air System vision system on the basis of a comparative, prospective, randomized against the reference method (sterile water + Betadine) during a gynecologic endoscopic surgery.

We propose to carry out a single-center, randomized, prospective trial comparing the efficacy in terms of reducing the number of cleaning FloShield Air System vision system, from a prospective, randomized during endoscopic surgery in gynecology.

After evaluation of the International Register of Clinical Trials Registry (https://clinicaltrials.gov/ct2/about-site) of the National Institutes of Health American no ongoing trial or released is interested or not interested at effectiveness of FloShield Air System vision device during endoscopic surgery in gynecology specifically on the primary endpoint.

Currently, the only Recruiting trial which concerns the system is entitled "Comparison FloShield Air System Versus clearify Visualization System (D-HELP)) (NCT02419911)." This is a non-academic comparative prospective trial efficiency.

The originality of our protocol resides in five points:

* His academic nature: the promoter is the University Hospital Tenon Hospital (AP-HP)
* It attempts to answer a clinical question frequently in clinical practice
* The feasibility: experience and surgical volume recruiting center in the endoscopic management should help support the computing power.
* Its safety for the patient
* The methodological basis helps support a level I evidence for this new material

ELIGIBILITY:
Inclusion Criteria:

Female or Male; 18 years of age or older; Patient scheduled for gynecologic paroscopic surgery under the care of the study investigator; Suitable candidate for surgery

Exclusion Criteria:

Unfit for surgery: concomitant disorders incompatible with the study or surgery (at the discretion of the investigator); Use of Surgiquest AirSeal®; Use of humidified insufflation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
number of Laparoscope removals during surgery | 0.5hr - 6hr

SECONDARY OUTCOMES:
medico economic cost effectiveness of the system | 0.5hr - 6hr
Evaluation of the quality of vision by the surgeon and his assistant end of the procedure using a visual analog scale | 0.5hr - 6hr

CONTACTS AND LOCATIONS:
Locations (1):
- Aphp, Tenon Hospital, Paris, Paris /france, France

REFERENCES:
- [Derived] Bendifallah S, Salakos E, Naoura I, Aristizabal P, Furet E, Zilberman S, Ballester M, Darai E. Prospective, randomized comparison of the use of FloShield Air System(R) versus the reference technique (water + povidone-iodine solution) during gynecologic endoscopic surgery to evaluate the operative lens vision quality. Surg Endosc. 2018 Mar;32(3):1593-1599. doi: 10.1007/s00464-017-5642-6. Epub 2017 Jun 22. PMID 28643058